CLINICAL TRIAL: NCT00294710
Title: A Twenty Six-week, Dose Titration Study to Evaluate the Efficacy and Safety of Aliskiren Compared to HCTZ With the Optional Addition of Amlodipine, Followed by a Second Twenty Six Weeks of Blinded Treatment, in Patients With Essential Hypertension
Brief Title: A Clinical Study to Compare Long-term Efficacy and Safety of an Aliskiren Based Regimen to a Hydrochlorothiazide Based Treatment Regimen With Optional Addition of Amlodipine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CSPP100A2323E
Record Dates: First submitted 2006-02-18; First posted 2006-02-22 (Estimated); Last update posted 2011-11-08 (Estimated); Status verified 2011-11

CONDITIONS: Hypertension
Keywords: Hypertension, aliskiren, hydrochlorothiazide, amlodipine
MeSH Terms: conditions — Hypertension | interventions — aliskiren

INTERVENTIONS:
Drug: Aliskiren

SUMMARY:
This study is designed to compare the long-term efficacy and safety of an aliskiren based regimen to an HCTZ based treatment regimen with optional addition of amlodipine in patients with essential hypertension

ELIGIBILITY:
Inclusion Criteria:

* Patients with essential hypertension

Exclusion Criteria:

* Severe hypertension
* History or evidence of a secondary form of hypertension
* History of myocardial infarction.
* Other protocol-defined inclusion exclusion criteria also apply.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 976 (Actual)
Dates: Start 2005-03; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in diastolic blood pressure after 52 weeks

SECONDARY OUTCOMES:
Change from baseline in systolic and diastolic blood pressure after 52 weeks
Diastolic blood pressure < 90 mmHg or a reduction of > 10 mmHg after 52 weeks
Achieve blood pressure control target of < 140/90 mmHg after 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Principal Investigator — Novartis Pharmaceuticals
Locations (2):
- Novartis, East Hanover, New Jersey, United States
- Investigative Centers, Germany

REFERENCES:
- [Derived] Schmieder RE, Philipp T, Guerediaga J, Gorostidi M, Smith B, Weissbach N, Maboudian M, Botha J, van Ingen H. Long-term antihypertensive efficacy and safety of the oral direct renin inhibitor aliskiren: a 12-month randomized, double-blind comparator trial with hydrochlorothiazide. Circulation. 2009 Jan 27;119(3):417-25. doi: 10.1161/CIRCULATIONAHA.107.750745. Epub 2009 Jan 12. PMID 19139391